CLINICAL TRIAL: NCT03672058
Title: Steps Ahead: Optimising Physical Activity and Health in Adults With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF UHL UL
Record Dates: First submitted 2018-09-03; First posted 2018-09-14 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis, CF
MeSH Terms: conditions — Cystic Fibrosis | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit plus personalised text messaging & Goal Setting (Experimental)
  Interventions: Other: Fitness tracker with goal setting and text message feedback
- Fitbit Only (Active Comparator)
  Interventions: Other: Fitness Tracker only

INTERVENTIONS:
Other: Fitness tracker with goal setting and text message feedback — Participants provided with a Fitbit and this will also be linked to Fitabase. The physiotherapist will discuss the participants' baseline physical activity levels and individual patient centred short and long-term goals will be set with each participant. Every week participants will be contacted via text message by their CF physiotherapist. The physiotherapist will review their online data and will provide feedback and encouragement on their progress. Goals will be reviewed for each participant.
  Arms: Fitbit plus personalised text messaging & Goal Setting
Other: Fitness Tracker only — Participants will be provided with the Fitbit and educated on how to use it. This will be linked to "Fitabase", an online monitoring system for data collection purposes, with the consent of the participants. However no goal setting will be completed and no feedback will be provided to the participants on their physical activity levels
  Arms: Fitbit Only

SUMMARY:
Physical activity is widely documented as one of the cornerstones of Cystic Fibrosis (CF) management as it is directly linked to mortality and quality of life. Levels of physical inactivity and sedentary behaviour have been poorly investigated among the CF population in Ireland. The measurement of these behaviours is important in order to monitor prevalence amongst people with CF (PWCF) and determine methods by which health care providers can assist with maintaining and enhancing physical activity.

The use of physical activity monitoring can provide health care providers with insightful real world analysis of physical activity and exercise behaviours. Over the last decade there has been many advancements in technology and fitness tracking with positive results being demonstrated in the healthy population and in chronic diseases such as Diabetes Mellitus II, post surgery and Multiple Sclerosis. Limited research has been conducted among PWCF to date.

The aim of this research project is to examine physical activity levels amongst PWCF and determine the effect of a 12 week randomised parallel intervention on a number of health outcomes.

Participants will be provided with an accelerometer to assess physical activity and sedentary behaviour at baseline. The participants will then undergo further baseline testing to determine exercise capacity, body composition, quality of life, breathlessness, sleep quality and wellbeing. Baseline short and long term goals will be established together with the participant and physiotherapist.

Participants will then be randomly allocated to either the intervention or the comparator. A researcher independent of the recruitment process (MC) will complete the first random allocation using a sealed opaque envelope. Following this a minimisation randomisation procedure will be completed based on lung function, where FEV1 of <70% predicted lung function will be classified as having mild lung disease. While those with an FEV1 of 30-50% predicted lung function will be classified as having moderate lung disease, with <30% indicating severe lung disease. Allocation will be revealed after recruitment and baseline assessments have occurred.

Both groups will receive a fitness tracker which will be linked to an online monitoring system (Fitabase) for 24 weeks.

The intervention group will receive personalised feedback via a text message every week on their physical activity levels as measured by their fitness tracker and progress on attainment of their goals established at the start of the study. Feedback will be provided from their CF physiotherapists.

The comparator group will not receive any feedback on their Fitbit data. After 12 weeks both groups will be re-assessed. Thereafter, both groups will continue with the Fitbits alone for 12 weeks. Finally outcome measures including lung function, physical activity levels, aerobic capacity, quality of life, sleep quality, muscle mass and well-being will be re-assessed again at 24 weeks.

Following the intervention semi structured interviews will be conducted to qualitatively establish satisfaction with the interventions and provide insight into barriers and enablers to achieving goals and physical activity levels.The results of this study may provide valuable insights into potential interventions to optimise the health and well-being of PWCF.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable CF patients
* Age > 18 years
* Confirmed diagnosis of CF
* Access to a smartphone/tablet to access and upload to Fitbit Application.
* Capacity and willingness to give explicit informed consent

Exclusion Criteria:

* FEV1 < 25%.
* Patients on the waiting list for lung transplantation and those who have undergone lung transplantation.
* Patients with an exacerbation in the four weeks prior to the study. For the purpose of this study pulmonary exacerbation will be defined as acute or subacute worsening of respiratory symptoms which warrant change in treatment (i.e., new oral or intravenous antibiotics). Patients can undergo testing once they are finished their antibiotics and deemed clinically stable.
* Patients dependent on supplemental oxygen for exercise.
* Pregnancy
* Participation in another clinical trial up to 4 weeks prior to the first baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Change in forced expiratory volume in 1 second (FEV1) (%predicted) | Baseline to 3 months and Baseline to 6 months
  Spirometry
Change in peak oxygen uptake (% predicted) | Baseline to 3 months and Baseline to 6 months
  Cardiopulmonary Exercise Testing
Change in number of steps per day | Baseline to 3 months and Baseline to 6 months
  Fitbit/Activpal

SECONDARY OUTCOMES:
Change in maximal aerobic power (%predicted) | Baseline to 3 months and Baseline to 6 months
  Cardiopulmonary Exercise Testing
Change in forced expiratory volume (FVC) (%predicted) | Baseline to 3 months and Baseline to 6 months
  Spirometry
Change in grip strength | Baseline to 3 months and Baseline to 6 months
  Hand Dynamometry
Change in body mass index (kg/m2) | Baseline to 3 months and Baseline to 6 months
  SECA Medical Body Composition Analyser
Change in muscle mass (kg) | Baseline to 3 months and Baseline to 6 months
  SECA Medical Body Composition Analyser
Change in percent body fat | Baseline to 3 months and Baseline to 6 months
  SECA Medical Body Composition Analyser
Change in Cystic Fibrosis Quality of Life Scale (CFQR) | Baseline to 3 months and Baseline to 6 months
  Measurement of the quality of life by the Cystic Fibrosis Questionnaire Revised (CFQ-R, Quality of life domains: Physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions. Symptom scales: Weight, respiratory, and digestion). There are 5 distinct 4-point Likert scale. Scores range from 0 to 100, with higher scores indicating better health.
Change in self reported physical activity (International Physical Activity Questionnaire Short Form) | Baseline to 3 months and Baseline to 6 months
  International Physical Activity Questionnaire. This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. It assesses 7 items to get a global score and then categorizes physical activity into low, moderate or high.
Pittsburgh Sleep Quality Index | Baseline to 3 months and Baseline to 6 months
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
The University of California San Diego (UCSD) Shortness of Breath Questionnaire | Baseline to 3 months and Baseline to 6 months
  To assess dyspnea associated with activities of daily living (ADLs). There are 24 items on this questionnaire. Each item is assessed on a 6-point scale (0 = "not at all" to 5 = "maximal or unable to do because of breathlessness"). Scores range from 0 to 120 with higher scores indicating activities of daily living are extremely limited by shortness of breath.
Change in wellbeing | Baseline to 3 months and Baseline to 6 months
  Alfred Wellness Score. This questionnaire assesses state of wellness to assist in providing best health care. There are 10 questions which are scored from 0-10. 10 reflects most well state of being possible while zero reflects least well state. Scores range from 0-100 with higher scores indicating good state of wellness.
Change in number of minutes spent in moderate to vigorous physical activity (MVPA) | Baseline to 3 months and Baseline to 6 months
  Fitbit/Activpal

OTHER OUTCOMES:
Time to exacerbation | Baseline to 3 months and Baseline to 6 months
Semi Structured Interviews | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roisin Cahalan, PhD, Principal Investigator — University of Limerick; Audrey Tierney, PhD, Principal Investigator — University of Limerick
Locations (1):
- University Hospital Limerick, Limerick, Ireland

REFERENCES:
- [Derived] Curran M, Tierney AC, Collins L, Kennedy L, McDonnell C, Jurascheck AJ, Sheikhi A, Walsh C, Button B, Galvin R, Casserly B, Cahalan R. Steps Ahead: optimising physical activity in adults with cystic fibrosis: Study Protocol for a pilot randomised trial using wearable technology, goal setting and text message feedback. HRB Open Res. 2020 Nov 16;3:21. doi: 10.12688/hrbopenres.13025.3. eCollection 2020. PMID 33283151